CLINICAL TRIAL: NCT01563146
Title: Assessing the Number of Rotavirus Related Hospitalizations in 11 Hospitals in Belgium - Season 2006-2007
Brief Title: Number of Rotavirus (RV) Related Hospitalizations in Belgium - Season 2006-2007
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116311
Record Dates: First submitted 2012-03-01; First posted 2012-03-26 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus; hospitals; Belgium
MeSH Terms: conditions — Rotavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Group A: All children ≤ 5 years old with a rotavirus detection test (inpatient and ambulatory tests) performed during the period of June the 1st 2006 and May the 31st 2007.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Each participating centre will be requested to generate a coded list of all stool samples taken during the study period (June 1st 2006- May 31st 2007) and analysed for rotavirus, in children aged ≤5 years.

SUMMARY:
This study aims to collect data and assess the number of rotavirus related hospitalizations in 11 hospitals in Belgium - season 2006-2007 in order to develop proper age-cohort analysis over time.

DETAILED DESCRIPTION:
This retrospective study will use anonymised data, extracted from hospital databases during the period of the 1st of June 2006 until the 31st of May 2007. IMS Health sales data will be used to provide rotavirus vaccine coverage estimates (Rotarix and Rotateq) for the Belgian population during the study period. Any additional source of vaccine coverage status describing rotavirus vaccine uptake in the study population will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Child aged ≤5 years;
* A stool sample has been provided for a rotavirus detection test during the study period;
* Laboratory test result of rotavirus is available.

Exclusion Criteria:

Not applicable.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged ≤5 years undergoing a RV detection test across 11 participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of the absolute number of rotavirus related hospitalisations in children up to five years old. | From June 1st 2006 up to 1 year

SECONDARY OUTCOMES:
Classification of patients with rotavirus hospitalisation by birth cohorts, gender, time of the event, vaccine coverage status. | From June 1st 2006 up to 1 year
Determination of the duration of rota-related hospitalisation for community acquired and nosocomial infection per birth cohort. | From June 1st 2006 up to 1 year
Evaluation of the herd effect. | From June 1st 2006 up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Standaert B, Strens D, Pereira P, Benninghoff B, Raes M. Lessons Learned from Long-Term Assessment of Rotavirus Vaccination in a High-Income Country: The Case of the Rotavirus Vaccine Belgium Impact Study (RotaBIS). Infect Dis Ther. 2020 Dec;9(4):967-980. doi: 10.1007/s40121-020-00345-y. Epub 2020 Oct 6. PMID 33025558
- [Derived] Standaert B, Strens D, Li X, Schecroun N, Raes M. The Sustained Rotavirus Vaccination Impact on Nosocomial Infection, Duration of Hospital Stay, and Age: The RotaBIS Study (2005-2012). Infect Dis Ther. 2016 Dec;5(4):509-524. doi: 10.1007/s40121-016-0131-0. Epub 2016 Oct 6. PMID 27714677
- [Derived] Standaert B, Strens D, Alwan A, Raes M. Medium- to Long-Term Impact of Rotavirus Vaccination on Hospital Care in Belgium: A 7-Year Follow-Up of the Rotavirus Belgium Impact Study (RotaBIS). Infect Dis Ther. 2016 Mar;5(1):31-44. doi: 10.1007/s40121-015-0099-1. Epub 2015 Dec 31. PMID 26721823